CLINICAL TRIAL: NCT06294964
Title: Sleep Education and Its Effects on Cardio-cerebrovascular Disease in Pudong Community Elderly Cohort
Brief Title: Intervention and Effect of Sleep Pattern on Cardio-cerebrovascular Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sleep Education
Record Dates: First submitted 2024-02-19; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases; Non-Communicable Chronic Diseases
Keywords: sleep intervention; sleep education; cardio-cerebrovascular diseases
MeSH Terms: conditions — Cardiovascular Diseases; Noncommunicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleep education group (Experimental)
  Interventions: Behavioral: sleep education, behavioral education
- routine management group (No Intervention)

INTERVENTIONS:
Behavioral: sleep education, behavioral education — Provide health education materials which covering sleep education, behavioral education, chronic diseases such as cardiovascular diseases. Topics touch on such as why you need healthy sleep? What methods can be used to regulate insomnia, and how to regulate sleep breathing problems? How do the elderly maintain a good sleep? What are the risk factors for cardiovascular and cerebrovascular diseases? How to reduce the risk of developing sleep disorders or chronic diseases through changing everyday life?
  Arms: sleep education group

SUMMARY:
Because of the growing population of older people, cardio-cerebrovascular diseases has been the most important aging-related chronic disease, studying the pathogenesis and early warning mechanisms of cardio-cerebrovascular diseases in depth, exploring optimal strategies for early diagnosis and treatments of cardio-cerebrovascular diseases has becoming the urgent public health problem in China. Aging causes cellular changes that change the sleep status in older adults, leading to an increased risk of disease and death. Meanwhile, the rising prevalence of chronic diseases among older adults also increases the impact of sleep deprivation. Insufficient sleep has being a serious challenge to the health status of the elderly. However, there is no clinically significant treatment for sleep disorders caused by chronic diseases. Medication helps to sleep but will also lead to drug dependence and increasing the risk of recurrent sleep disorders, which is unfavorable for disease control.

Studies have shown that older adults who sleep 7-8 hours at night have better physical and mental health, cognition and quality of life. Shorter sleep durations (6 hours or less) and longer sleep durations (greater than 9 hours) had strong associations with adverse health outcomes such as cardiovascular, metabolic, immune, cognitive diseases, other psychiatric disorders, and mortality.

Therefore, on the basis of the established Pudong community cohort, the project applicant led the team to adopt an open-label, blind endpoint, and cluster-randomized two-phase trial method to randomly assign cohort members into intervention group and control group. According to the sleep health intervention plan formulated by the clinical team, family doctor provides health education materials according to the actual situation of the intervention group regularly. Family doctors in the control group used conventional management methods. The final assessment was that compared to control group, whether the intervention group improved members' sleep quality, reduced members' cardiovascular disease events, and individual cardiovascular disease morbidity and all-cause mortality during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥ 60 years；
* Participate in the cohort of Shanghai Pudong community;
* There is a family doctor or regular family doctor in the neighborhood committee who is willing to participate in this project；
* Sign the informed consent;
* No immigrant intention in the next 3 years;
* Not pregnant or planning to become pregnant;
* No malignant tumor, life expectancy ≥ 3 years;
* Participating in the annual community-based elderly group examination project in the next three years

Exclusion Criteria:

* Those who are unwilling to participate in clinical research;
* Patients who participate in other clinical research;
* Patients with a history of severe mental illness or deafness;
* Patients who cannot complete follow-up

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12800 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
the incidence and/or prevalence of cardiovascular diseases such as myocardial infarction, stroke, heart failure, and cardiovascular death | 3 years
  the incidence and/or prevalence of cardiovascular diseases such as myocardial infarction, stroke, heart failure, and cardiovascular death

SECONDARY OUTCOMES:
all cause death | 3 years
  all cause death

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, MD, PhD, Principal Investigator — Cardiology, Ren Ji Hospital, Shanghai, China
Locations (1):
- Cardiology, Ren Ji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No